CLINICAL TRIAL: NCT03689881
Title: Value of Tomosynthesis for Detection of Sacro-iliitis: a Prospective Comparative Study
Brief Title: Value of Tomosynthesis for the Detection of Sacro-iliitis (TOMOS SI)
Acronym: TOMOS SI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: DMS Apelem (Industry); Thales (Unknown); Digisens (Unknown); Medecom (Unknown); BPIfrance (Other); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0328
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2018-09

CONDITIONS: Sacroiliitis
Keywords: Sacroiliitis; SI joint; tomosynthesis; CT; Xray
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tomosynthesis (Experimental): Tomosynthesis of SI joints
  Interventions: Device: Tomosynthesis of SI joints

INTERVENTIONS:
Device: Tomosynthesis of SI joints — All patients will undergo additional tomosynthesis performed per study protocol along with Xray and CT performed as part of standard imaging evaluation of sacroillitis.
  Tomosynthesis of SI joints will be performed on a digital Tomosynthesis system (PLATINUM dRF v2 DMS/APELEM), with a single acquisition followed by coronal image reconstruction.

SUMMARY:
Spondyloarthropathies (SpAs) are chronic inflammatory diseases encompassing ankylosing spondylitis, psoriatic arthritis, reactive arthritis, enteropathic arthropathy, and undifferentiated SpA.

In 2001, the estimated prevalence of SpA was 1.5% worldwide. Sacroiliitis is a condition caused by inflammation within the sacroiliac joint. It is the most frequent damage of SpA depicted at imaging evaluation.

Conventional radiography (X-ray) is usually used to depict the structural changes associated with sacroiliitis.

However further evaluation often requires additionnal computed tomography (CT).

Tomosynthesis is an Xray-based imaging technology which allows reconstruction of multiple section images from a set of projection images acquired as the x-ray tube moves along a prescribed path. The advantagee of tomosynthesis is the significant reduction of radiation dose exposure compared to CT Tomosynthesis is currently used in the field of breast imaging and pneumology. Very few studies have examined the value of tomosynthesis for osteoarticular imaging.

The study aims at evaluating the diagnostic performances of tomosynthesis as compared to standard X-ray and CT, in patients with a clinical suspicion of sacroiliitis.

the investigators hypothesize that tomosynthesis is superior to conventional radiography for detection of sacroiliitis and is at least equal to CT with lower irradiation.

DETAILED DESCRIPTION:
Consecutive patients referred to CT for exploration of sacrollitis will be included and investigated with standard radiography, CT and tomosynthesis of SI joints.

Imaging examinations will be performed at day of enrollment as follow : X-ray and CT as standard management and tomosynthesis as additional evaluation. CT will be considered as the reference standard Sacroiliitis will be assessed in a centralized, blind and randomized retrospective reading of all imaging modalities by two independent radiologists.

Diagnostic performances and radiation doses of tomosynthesis will be compared to those of standard CT and X-ray examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over referred for suspected sacroiliitis.
* Patients who have entered into their participation agreement by signing the informed consent form.
* Patient affiliated to a social security scheme or beneficiary.

Exclusion Criteria:

* Pregnant or lactating women.
* Vulnerable people according.
* Major people placed under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of bone erosions and other structural lesions of SI joints | 1 day of enrollment
  sacroiliitis will be assessed independently for each imaging modality according to the modified New York criteria

SECONDARY OUTCOMES:
radiation dose | 1 day of enrollment
  Radiation dose will be measured for each imaging evaluation and calculated as the effective dose in millisievert (mSv).
inter reader agreement for the evaluation of sacroiliitis at tomosynthesis | at the end of patients enrollment
  Inter reader agreement will be measured at retrospective evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cyteval, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Imaging department- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No